CLINICAL TRIAL: NCT04356118
Title: Efficacy and Safety of Recombinant Human Endostatin in Non-Small Cell Lung Cancer With Leptomeningeal Metastasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hui Bu (Other)
Responsible Party: Sponsor-Investigator, Hui Bu, Study Principal Investigator, Hebei Medical University
Organization: Hebei Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH 005
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Leptomeningeal Metastasis
Keywords: Recombinant Human Endostatin; Non-Small Cell Lung Cancer with Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Endostatins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endostatin Therapy for NSCLC of LM (Experimental): Recombinant Human Endostatin + intrathcal methotrexate+Targeted drugs for non-small cell lung cancer
  Recombinant Human Endostatin:15mg/endostatin;The dose is 7.5mg/㎡/d，Once a day for two weeks, take a week off,start the next cycle, up to four cycles.
  intrathcal methotrexate :Intrathecal chemotherapy specified dose on specified days.
  Targeted drugs for non-small cell lung cancer:
  EGFR Mutation: Erlotinib，Afatinib，Osimertinib, et al. ALK ROS1 Mutation:Crizotinib,Ceritinib,Alectinib ,et al. BARF Mutation:Vemurafenib,et al. Other Mutation: other Targeted drugs .
  Interventions: Drug: Recombinant Human Endostatin; Drug: intrathcal methotrexate; Drug: Targeted drugs for non-small cell lung cancer

INTERVENTIONS:
Drug: Recombinant Human Endostatin — endostatin 7.5mg/㎡/d，Once a day for two weeks, take a week off,start the next cycle, up to four cycles .We advocate a highly individualized treatment plan according to each patients specific manifestations of the disease process.
  Other Names: Endostatin
Drug: intrathcal methotrexate — Intrathecal chemotherapy specified dose on specified days.
Drug: Targeted drugs for non-small cell lung cancer — EGFR Mutation: Erlotinib，Afatinib，Osimertinib, et al. ALK ROS1 Mutation:Crizotinib,Ceritinib,Alectinib ,et al. BARF Mutation:Vemurafenib,et al. Other Mutation: other Targeted drugs .

SUMMARY:
The purpose of this study is to observe the clinical effect and safety of Recombinant Human Endostatin in non-small cell lung cancer with leptomeningeal metastasis

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old
2. Pathologically proven non-small cell lung cancer
3. Karnofsky performance status ≥ 40
4. LM diagnosis was based on the detection of malignant cells in the CSF, the focal or diffuse enhancement of leptomeninges, and nerve roots or the ependymal surface on gadolinium-enhanced MRI .
5. No severe abnormal liver and kidney function;
6. Patients have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Evidence of bleeding diathesis or serious infection
2. Serious cardiovascular disease (congestive heart failure, uncontrollable arrhythmia, unstable angina, myocardial infarction, serious heart valve disease, resistant hypertension)
3. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Leptomeningeal Metastasis Overall survival | 36 months
  Leptomeningeal Metastasis Overall survival defined as time from LM diagnosis to death due to any cause or last follow-up
Neurological Progression Free Survival | 36 months
  From the start of treatment until central nervous system metastase progression or death due to any cause
The incidence of adverse reactions | 36 months
  From date of first dose up to assessed from April 2020 to April 2023 (In accordance with the standard of CTCAE)

SECONDARY OUTCOMES:
Objective Response Rate | 36 months
  ORR, proportion of patients with a best overall response of complete response or partial response (CR+PR)
Neurological assessment | 36 months
  In accordance with the standard of Response Assessment in Neuro-Oncology(RANO) Neurological Assessment group.The maximum value is 29 and the minimum value is 0.The higher scores mean a worse outcome.
progression-free survival | 36 months
  Proportion of patients progression-free by investigator assessment per RECIST v1.1
Overall survival | 36 months
  defined as time from Non-Small Cell Lung Cancer diagnosis to death due to any cause or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hui Bu, Principal Investigator — The Second Hospital of Hebei Medical University